CLINICAL TRIAL: NCT03777956
Title: The Effect of Lacosamide in Peripheral Neuropathic Pain: a Randomized, Double-blind, Placebo Controlled, Phenotype-stratified Study
Brief Title: The Effect of Lacosamide in Peripheral Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID 19 and recruitment problems
Sponsor: Danish Pain Research Center (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LACOSAMIDE-2018; 2018-003110-40 (EudraCT Number)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain; Neuropathy;Peripheral; Neuropathy, Painful; Neuropathy, Diabetic; Neuropathy
MeSH Terms: conditions — Neuralgia; Neuritis; Neuropathy, Painful; Diabetic Neuropathies | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacosamide (Active Comparator): Lacosamide (50 mg) are given as capsules and taken orally twice a day, up to 200 mg b.i.d.
  Interventions: Drug: Lacosamide
- Placebo (Placebo Comparator): Placebo are given as capsules, same as lacosamide, and taken orally twice a day, without active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacosamide — Lacosamide (50 mg) and identical placebo are given as capsules and taken orally twice a day, up to 200 mg b.i.d.
  Arms: Lacosamide
Drug: Placebo — Identical placebo are given as capsules and taken orally twice a day.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to compare the change in pain intensity during treatment with a sodium-channel blocker (lacosamide) in patients with peripheral neuropathic pain with and without the irritable nociceptor phenotype.

DETAILED DESCRIPTION:
The main purpose of this study is to compare the change in pain intensity during treatment with a sodium-channel blocker (lacosamide) in patients with peripheral neuropathic pain with and without the irritable nociceptor phenotype. As this is a mechanistic study, the main purpose is to compare the change in pain intensity in patients who receive an expected sufficiently effective dose of lacosamide. As supportive evidence for a drug-specific predictive biomarker, the purpose is also to compare the change in pain intensity during lacosamide vs. placebo for the two phenotypes.

We hypothesize that the sodium-channel blocker lacosamide will be more effective in patients with the irritable nociceptor than those without the non-irritable nociceptor phenotype, and that lacosamide is more effective than placebo in patients with the irritable nociceptor phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Probable or definite peripheral neuropathic pain for at least 3 months (Finnerup et al. 2016)
3. Average pain intensity of at least 4 and not above 9 on a 0-10 NRS during the 7-day baseline week (Dworkin et al. 2012).
4. Written informed consent.

Exclusion Criteria:

1. Other causes of pain in the same area, or other concomitant pain that cannot be distinguished from the neuropathic pain
2. Patient who cannot cooperate or are unable to complete the project and patients who do not speak Danish.
3. Known and current cardiac conduction disturbance (2⁰ or 3⁰ atrioventricular (AV) block, prolonged QTc interval > 450 ms, heart rate <50 or >110 bpm, a QRS interval >120ms (ECG required)), significant cardiac, renal or liver disease or other severe illness. In patients treated with pregabalin also PQ interval > 0,2s and cardiac disease. Sitting diastolic blood pressure below 50 mmHg or above 105 mmHg.
4. Major depressive episode within 6 months, recurrent depressive disorder or other significant psychiatric disease, alcohol, illicit drug or drug abuse.
5. Pregnancy or lactation
6. Woman of childbearing potential, unless they use and acceptable effective contraception measure as defined in the Clinical Trials Facilitation Group (CTFG) during the study and at least 2 weeks after, or if their male partner is vasectomized and their sole partners. Negative pregnancy test is required.
7. Known allergy to lacosamide or excipients.
8. Concomitant pain treatment with tricyclic antidepressants, topical analgesics (lidocaine, capsaicin), lamotrigine, oxcarbazepine, cannabinoids or strong opioids that cannot be discontinued. Other treatment for neuropathic pain are allowed in a stable dose (from 14 days before randomization to completion of the trial), if they cannot be tapered off completely.
9. Concomitant treatment with products known to be associated with PQ (PR) prolongation other than pregabalin.
10. Patients inappropriate for placebo
11. Planned surgery
12. Use of sodium channel blockers within at least five half-lives and investigational drugs within 30 days.
13. Patients on controlled sodium diet, unless the amount of sodium in the capsules is acceptable for their diet.
14. The score "yes" on item 4 or item 5 of the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS), if the ideation occurred in the past 6 months, or "yes on any item of the Suicidal Behaviour section, except for the "Non-suicidal Self Injurious Behaviour" if this behaviour occurred in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 12 weeks
  The difference in the mean value of the patient's daily ratings of average pain intensity in the baseline week and the last week during treatment as experienced during the past 24 hours rated on a 0-10 point numeric rating scale (NRS; 0 = no pain, 10 = worst possible pain).
  The primary objective is to compare the change in pain intensity from baseline to last week of lacosamide treatment in patients with and without the irritable nociceptor phenotype in the PP population.
  The supportive objective is to compare the effect of lacosamide vs. placebo in the two phenotype groups in the PP population. Although we do not expect a phenotype difference in the response to placebo, a comparison of the effect of lacosamide vs. placebo is needed to justify that the phenotype is a predictive biomarker for the effect of lacosamide.

SECONDARY OUTCOMES:
Pain relief | 12 weeks
  (complete, good, moderate, mild, none, worse pain) . Measured at last visit/end of treatment period.
Use of escape medicine (paracetamol) during treatment period. | 12 weeks
  Number of paracetamol tablets during the 12 weeks treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna B Finnerup, Professor, Study Director — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Background] Dworkin RH, Turk DC, Peirce-Sandner S, Burke LB, Farrar JT, Gilron I, Jensen MP, Katz NP, Raja SN, Rappaport BA, Rowbotham MC, Backonja MM, Baron R, Bellamy N, Bhagwagar Z, Costello A, Cowan P, Fang WC, Hertz S, Jay GW, Junor R, Kerns RD, Kerwin R, Kopecky EA, Lissin D, Malamut R, Markman JD, McDermott MP, Munera C, Porter L, Rauschkolb C, Rice ASC, Sampaio C, Skljarevski V, Sommerville K, Stacey BR, Steigerwald I, Tobias J, Trentacosti AM, Wasan AD, Wells GA, Williams J, Witter J, Ziegler D. Considerations for improving assay sensitivity in chronic pain clinical trials: IMMPACT recommendations. Pain. 2012 Jun;153(6):1148-1158. doi: 10.1016/j.pain.2012.03.003. Epub 2012 Apr 9. PMID 22494920
- [Derived] Carmland ME, Kreutzfeldt M, Holbech JV, Andersen NT, Jensen TS, Bach FW, Sindrup SH, Finnerup NB. Effect of lacosamide in peripheral neuropathic pain: study protocol for a randomized, placebo-controlled, phenotype-stratified trial. Trials. 2019 Oct 11;20(1):588. doi: 10.1186/s13063-019-3695-7. PMID 31604475